CLINICAL TRIAL: NCT04265781
Title: Phase 1 Dose Escalation Study to Investigate Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses of BAY 1817080 in Japanese Healthy Adult Male Participants in a Single-center, Randomized, Single-blind, Placebo-controlled Design
Brief Title: Study on the Safety of Drug BAY1817080 at Different Doses and the Way the Body Absorbs and Eliminates the Drug in Japanese Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: 19738
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Endometriosis Related Pain; Overactive Bladder; Diabetic Neuropathic Pain; Refractory or Unexplained Chronic Cough
Keywords: Refractory or unexplained chronic cough; Healthy volunteers; P2X3 receptor antagonist
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose escalation BAY1817080 (Experimental): Participants receive dose 1 to 3 of BAY1817080 as a single dose on Day 1.
  Interventions: Drug: BAY1817080
- Dose expansion BAY1817080 (Experimental): Participants receive the highest dose 3 of BAY1817080 twice daily (BID) from Day 1 until Day 13 and a single dose on Day 14.
  Interventions: Drug: BAY1817080
- Dose escalation Placebo (Placebo Comparator): Participants receive placebo tablets orally as a single dose on Day 1.
  Interventions: Drug: Matching Placebo
- Dose expansion Placebo (Placebo Comparator): Participants receive placebo tablets as BID multiple doses from Day 1 until Day 13 and as a single dose on Day 14.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: BAY1817080 — Three different doses over the course of study
  Arms: Dose escalation BAY1817080; Dose expansion BAY1817080
Drug: Matching Placebo — Matching Placebo to BAY1817080
  Arms: Dose escalation Placebo; Dose expansion Placebo

SUMMARY:
Researchers in this study want to learn about the safety of drug BAY1817080 at different doses and the resulting blood levels of the study drug in Japanese healthy adult male participants. Study drug BAY1817080 is a drug under development with a goal to suppress pain and chronic cough. It works by binding to and blocking proteins expressed on the sensory nerves of the womb tissue, bladder or airway which are oversensitive in the patients with endometriosis (a condition where the tissue that usually grows inside the womb grows outside of the womb), overactive bladder (a condition that causes a sudden urge to urinate often or more frequently) and long-standing cough with or without clear causes.

Participants in this study will receive either the study drug or placebo tablets (a placebo looks like the test drug but does not have any medicine in it). The dosage will be either one single dose of study drug/placebo received on only one day or multiple doses of study drug/placebo received twice daily for 13 days plus one dose in the morning of the 14th day. The total study duration for each participant will be usually no more than 42 days. Blood samples will be collected from the participants to monitor the safety and measure the blood level of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 20 to 45 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs, laboratory tests, and ECG.
* Non-smoker for at least 6 months and with a pack year history of equal to or less than 5 years
* Race: Japanese.
* BMI: above or equal 18.0 and below or equal 30.0 kg/m² at the screening visit.
* Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Men of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period between signing of the ICF and 90 days after the last administration of study intervention.

Exclusion Criteria:

* Any findings from the medical examination (including medical history, physical examination, vital signs, laboratory tests and ECG) deviating from normal and deemed by the investigator to be of clinical relevance
* Relevant diseases potentially interfering with the study objectives within the 4 weeks before screening or between screening and randomization
* Any febrile illness within the four weeks before screening or between screening and randomization
* Any known presence or history of severe allergies, non-allergic drug reactions, or multiple drug allergies
* Known or suspected malignant tumors or carcinoma in situ
* Any history of malignant tumors
* Any known or suspected benign tumors of the liver and/or pituitary gland
* Known liver disease: existing acute or chronic progressive liver disease, e.g. disturbance of bilirubin excretion (Dubin-Johnson and Rotor syndromes); disturbances of bile secretion and flow (cholestasis); presence or history of liver tumors (benign or malignant). Note: According to this criterion there must have been an interval of at least 6 months between the subsidence of any viral hepatitis (normalization of liver parameters) and the screening visit.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events (TEAE) after single dose of BAY1817080 | Up to 14 days
Severity of treatment-emergent adverse events after single dose of BAY1817080 | Up to 14 days
Frequency of treatment-emergent adverse events after multiple doses of BAY1817080 | Up to 27 days
Severity of treatment-emergent adverse events after multiple doses of BAY1817080 | Up to 27 days

SECONDARY OUTCOMES:
Maximum plasma concentration of BAY1817080 after single dose (Cmax) | At 0 hour before study drug administration and up to 15 hours after study drug administration at Day 1 and at 0 hours on Day 2 to Day 10
Area under the concentration-time curve of BAY1817080 after single dose (AUC) | At 0 hour before study drug administration and up to 15 hours after study drug administration at Day 1 and at 0 hours on Day 2 to Day 10
  In the case of extrapolated portion of AUC exceeding20% [%AUC(tlast-∞) >20%], the parameter AUC(0-tlast) may be evaluated as main parameter
Maximum plasma concentration of BAY1817080 after multiple doses (Cmax,md) | At 0 hours before drug administration and up to 12 hours after drug administration on Day 1, at 0 hours from Day 2 to Day 9 and from Day 11 to Day 12, at 0 and 12 hours on Day 13, at 0 hours until 15 hours on Day 14, and at 0 hours from Day 15 to Day 23
Area under the concentration-time curve of BAY1817080 after multiple dose (AUCτ,md) | At 0 hours before drug administration and up to 12 hours after drug administration on Day 1, at 0 hours from Day 2 to Day 9 and from Day 11 to Day 12, at 0 and 12 hours on Day 13, at 0 hours until 15 hours on Day 14, and at 0 hours from Day 15 to Day 23

CONTACTS AND LOCATIONS:
Locations (1):
- Hakata Clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share data. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Li X, Haranaka M, Li H, Liu P, Chen H, Klein S, Reif S, Francke K, Friedrich C, Okumura K. P2X3 Receptor Antagonist Eliapixant in Phase I Clinical Trials: Safety and Inter-ethnic Comparison of Pharmacokinetics in Healthy Chinese and Japanese Participants. Clin Pharmacokinet. 2024 Jun;63(6):901-915. doi: 10.1007/s40262-024-01387-y. Epub 2024 Jun 21. PMID 38907175
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/